CLINICAL TRIAL: NCT06702501
Title: Minimally Invasive Pericardiotomy as a New Treatment for Heart Failure With Preserved Ejection Fraction - The PeriCut Catheter System Early Feasibility Study (REIMAGINE HFpEF)
Brief Title: The PeriCut Catheter System Early Feasibility Study (REIMAGINE-HFpEF)
Acronym: REIMAGINE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Failure Solutions, Inc. (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL00001
Record Dates: First submitted 2024-10-30; First posted 2024-11-25 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure Solutions; Heart Failure with Preserved Ejection Fraction; PeriCut; Pericardiotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single Arm - Procedure & Follow up (Experimental): Subjects will undergo minimally invasive pericardiotomy under fluoroscopic guidance and general anesthesia using the PeriCut Catheter System
  Interventions: Device: PeriCut Catheter System performs minimally invasive pericardiotomy

INTERVENTIONS:
Device: PeriCut Catheter System performs minimally invasive pericardiotomy — The PeriCut Catheter System will incise the pericardium to reduce filling pressures of the heart.

SUMMARY:
The PeriCut early feasibility study will evaluate the safety and feasibility of successfully performing a minimally invasive pericardiotomy in patients with heart failure with preserved ejection fraction using the PeriCut Catheter System.

DETAILED DESCRIPTION:
The PeriCut EFS is a non-randomized, open label, multi-site study testing a new minimally invasive pericardiotomy device for the treatment of heart failure with preserved ejection fraction (HFpEF).

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 30 years
* Symptoms of severe dyspnea (NYHA Class III-IV) without evidence of a non-cardiac or ischemic explanation for dyspnea
* Ejection fraction of ≥50%, determined on most recent imaging study within the preceding 2 years (730 days), with no change in clinical status, suggesting potential for deterioration in systolic function.
* Documentation history of at least one of the following:

Any previous hospitalization for HF (>30 days prior to enrollment) with radiographic evidence of pulmonary congestion (pulmonary venous hypertension, vascular congestion, interstitial edema, pleural effusion) or Elevated NT-proBNP (>300 pg/ml or >600 pg/ml if in atrial fibrillation) or Echocardiographic evidence of diastolic dysfunction/elevated filling pressures manifested by medial E/e' ratio ≥15 and/or left atrial enlargement and chronic treatment with a diuretic for signs or symptoms of heart failure or Historical catheterization documented elevated filling pressures at rest (PCWP ≥15 or LVEDP ≥18) or with exercise (PCWP ≥25), prior to consent.

* Catheterization documented elevated filling pressures at rest (PCWP ≥15 or LVEDP ≥18) or with exercise (PCWP ≥25) during the screening/baseline visit (after consent)
* Ambulatory with ability to complete 6-minute walk and cardiopulmonary exercise test (not wheelchair / scooter dependent)

Exclusion Criteria

* Recent (< 30 days) hospitalization for heart failure
* Left (> 6 cm) ventricular dilation noted on cardiac imaging study (echocardiography or MRI) within 6 months prior to enrollment.
* Any hemoglobin (Hgb) < 8.0 g/dl within 30 days prior to enrollment
* Any GFR < 20 ml/min/1.73 m2 within 30 days prior to enrollment
* Significant alternative cause of dyspnea such as severe chronic obstructive pulmonary disease or ischemia that is a primary contributor to symptoms, in the opinion of the Investigator.
* Myocardial infarction (MI), unstable angina, catheter ablation for atrial fibrillation, biventricular pacing device implant, or percutaneous coronary intervention (PCI) within 90 days prior to enrollment
* Any prior cardiac surgery
* Documented stroke, CVA, TIA, deep vein thrombosis, pulmonary emboli, or suspected neurological event within 180 days prior to enrollment
* Diagnosis of obstructive hypertrophic cardiomyopathy
* Known infiltrative cardiomyopathy (e.g., amyloid)
* Known pericardial disease (constriction, pericarditis, tamponade)
* Known allergy or sensitivity to contrast media that cannot be adequately pre-treated prior to the procedure.
* Active myocarditis
* Significant congenital anomaly, anatomic, or comorbid medical problem that, in the opinion of the Investigator, would preclude enrollment in the study.

Active collagen vascular disease

* Significant valvular heart disease (greater than mild stenosis or greater than moderate regurgitant lesions)
* Acute or chronic severe liver disease, as evidenced by any of the following: encephalopathy, variceal bleeding, INR > 1.7 in the absence of anticoagulation treatment.
* Untreated severe obstructive sleep apnea (if known)
* Implantation or planned implantation of any left atrial shunts or implantable devices used to treat heart failure.
* Terminal illness (other than HF) with expected survival of less than 1 year
* Enrollment or planned enrollment in another therapeutic clinical trial in the next 6 months.
* Inability to comply with planned study procedures or follow-up requirements, including cardiac MRI (e.g., claustrophobia or absolute contraindication to MRI)
* Women who are currently pregnant, plan to become pregnant, or are currently breastfeeding.
* Intolerance or contraindication to colchicine

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Safety | 30 day follow up
  Characterize the incidence of serious device and procedure related safety events at 30 days post procedure
Assessment of Acute Procedural Success | 30 day follow up
  Characterize the rate of acute treatment success of the PeriCut Catheter System to complete the pericardiotomy procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Barry Borlaug, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Corporate Website — http://www.heartfailureinc.com